CLINICAL TRIAL: NCT04667130
Title: Preventive Complex Program for Newly Diagnosed People With Multiple Sclerosis
Brief Title: Preventive Program in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamila Řasová (Other)
Responsible Party: Sponsor-Investigator, Kamila Řasová, associate professor PhDr. Kamila Řasová, Ph.D., Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EK-VP/25/0/2014
Record Dates: First submitted 2020-11-20; First posted 2020-12-14 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
Keywords: Preventive program; Multiple Sclerosis; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preventive Complex Program for Newly Diagnosed People With Multiple Sclerosis (Experimental): Providing information about the possibilities of physiotherapy, Computer Kinesiology, psychotherapy, Motor progam activating therapy, aerobic exercise
  Interventions: Behavioral: Preventive Complex Program for Newly Diagnosed People With Multiple Sclerosis

INTERVENTIONS:
Behavioral: Preventive Complex Program for Newly Diagnosed People With Multiple Sclerosis — Preventive program included informations of the possibilities of physiotherapy in the treatment of multiple sclerosis focused on fatigue management - recommending lifestyle changes. Program included a the treatment of psychosomatic, viscerosomatic functional disorders by reflexively poor connection through the locomotor system using computer kinesiology, psychotherapy, manual therapy - where patients are corrected into a postural position and the joints are functionally centred, and aerobic exercise to influence fatigue and improve the performance of the cardiovascular system.

SUMMARY:
This study monitor the immediate and persistent impact of a preventive complex six-month program specifically developed for newly diagnosed people with multiple sclerosis on fatigue, mental and physical fitness, and quality of life. The study determined whether changes in clinical function are related to changes in neurohormones, and whether the effect of therapy is dependent on the active approach of study participants.

DETAILED DESCRIPTION:
The patients who were newly diagnosed with MS underwent a six-month preventive comprehensive program, which included individual physiotherapy focused on the treatment of functional disorders of the loco-motor system and therapy on a neurophysiological basis, group psychotherapy and controlled aerobic training. The participants were examined three times - before the start of the physiotherapy program, immediately after its completion and six months apart. Influence on physical fitness (spiroergometric examination), fatigue (Modify Fatigue Impact Scale, fatigue scale for motor and cognitive functions), depression (Beck scale for evaluation of depression), admission of disease RS (Inventory of admission of multiple sclerosis, quality of life) life and selected neurohormones (dehydroepiandrosterone-DHEA, dehydroepiandrosterone sulphate - DHEAS, cortisol).

ELIGIBILITY:
Inclusion Criteria:

* definite MS
* stable clinical status in the preceding 3 months
* imumnomodulatory treatment for at least two years (including glatiramer acetate, interferon beta-1a, 1b, mitoxantrone, fingolimod, natalizumab)
* Expanded Disability Status Scale (EDSS)≤6
* predominant motor impartment
* six months or more without any physiotherapy
* ability to undergo ambulatory physiotherapy

Exclusion Criteria:

* other neurological disease or conditions disabling movement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Questionnaires - The Fatigue scale for motor and cognitive functions | change after six months of the program and after next six moths without therapy is being assessed
  FSMC - is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue).
Questionnaires - The Satisfaction With Life Scale | change after six months of the program and after next six moths without therapy is being assessed
  The scale measures the current level of satisfaction with one's own life. Investigators express the extent to which they agree or disagree with the five statements. The rating scale contains 7 points (1- "strongly disagree" and 7 - "strongly agree"). The maximum number of points on the scale is 35 (maximum satisfaction with your life) and the minimum number of points is 5 (dissatisfaction with your life).
Questionnaires - Multiple Sclerosis Acceptance Questionnaire | change after six months of the program and after next six moths without therapy is being assessed
  This questionnaire consists of 20 statements that relate to the lives of patients with MS. The rating scale has seven points (1- "never pays" to 7 - "always pays"). The minimum value is 20 (minimum adaptation to the diagnosis of MS for a large limitation of the normal life of MS) and the maximum value is 140 points (maximum adaptation to the diagnosis of MS - without the limitation of the normal life of MS) .
Questionnaires - Beck Depression Inventory Score | change after six months of the program and after next six moths without therapy is being assessed
  questionnaire is divided into thirteen categories and patients select a statement in each category which best fits their current feelings on the scale ranged from 0 (the best feelings) to 3 (the worst feelings). The maximum value of the total scale is 39 and shows the worst feeling of the person.

SECONDARY OUTCOMES:
Ventilation capacity | change after six months of the program and after next six moths without therapy is being assessed
  Forced vital capacity = FVC [ l ]
Metabolic utilization | change after six months of the program and after next six moths without therapy is being assessed
  maximal muscle performance = Rmax [ Watt kg-1 ]
Maximal oxygen uptake | change after six months of the program and after next six moths without therapy is being assessed
  VO2 kg-1 [ VO2max.kg-1 ]
Maximal oxygen pulse | change after six months of the program and after next six moths without therapy is being assessed
  VO2 HR-1 kg-1 [ VO2max.TF-1 ]
Relative ventilation | change after six months of the program and after next six moths without therapy is being assessed
  [ VEmax.kg-1 ]
Cortisol | change after six months of the program and after next six moths without therapy is being assessed
  levels of cortisol [ ng/mL ]
Cortizone | change after six months of the program and after next six moths without therapy is being assessed
  levels of cortisone[ ng/mL ]
Dehydroepiandrosterone (DHEA) | change after six months of the program and after next six moths without therapy is being assessed
  levels of DHEA [ ng/mL ]
7β-hydroxydehydroepiandrosterone (7β-OH-DHEA ) | change after six months of the program and after next six moths without therapy is being assessed
  levels of 7β-OH-DHEA [ ng/mL ]
7-oxo dehydroepiandrosterone (7-oxo-DHEA ) | change after six months of the program and after next six moths without therapy is being assessed
  levels of 7-oxo-DHEA [ ng/mL ]

OTHER OUTCOMES:
Questionnaires - Modified Fatigue Impact Scale | change after six months of the program and after next six moths without therapy is being assessed
  This scale consists of 21 statements that describe how often fatigue has affected a person during last four weeks. Each statement is ranged from 0 (never) to 4 (almost, always). The maximum value of the scale is 84.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, Ph.D., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Kamila Řasová, Prague, Czechia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04667130/Prot_SAP_ICF_000.pdf